CLINICAL TRIAL: NCT02228551
Title: Augmented Renal Clearance in the Adult Non-critically Ill Surgery Patient: a Prospective Point Prevalance Study and Identification of Risk Factors
Brief Title: Augmented Renal Clearance in the Adult Non-critically Ill Surgery Patient: a Prospective Point Prevalance Study
Acronym: ARCPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S55822-S55712
Record Dates: First submitted 2014-07-18; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2013-11

CONDITIONS: Prevalence of Augmented Renal Clearance; Risk Factors for Augmented Renal Clearance
Keywords: Augmented renal clearance; non-critically ill; surgery; prevalence; risk factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARC PPS (Other): Augmented renal clearance Point prevalence study
  Interventions: Other: Augmented renal clearance Point prevalence study

INTERVENTIONS:
Other: Augmented renal clearance Point prevalence study — An 8-hour urine collection was carried out to determine the CrCl8h. Participants were asked to empty the bladder at the start of the collection. From then, patients were asked to collect urine in a recipient during the following 8 hours. If an indwelling transurethral or suprapubic urinary catheter was in situ, the collection bag was emptied at the start of the collection. After 8 hours, total urinary volumes (Uv8h) were measured with a measuring cup and urinary creatinine concentrations were determined by laboratory analysis. Midterm serum creatinine samples were obtained at 4 hours after the start of the urinary collection. Based on these values, CrCl8h was calculated according to the standard formulas and normalized to a body surface area (BSA) of 1.73m².

SUMMARY:
This point prevalence study investigates the prevalence of augmented renal clearance (i.e. a measured 8-hour urinary creatinine clearance >= 120 ml/min/1.73m²) in an adult non-critically ill abdominal and trauma surgery population. Secondary objectives are the identification of risk factors associated with ARC in this specific study population.

DETAILED DESCRIPTION:
This point prevalence study investigates the prevalence of augmented renal clearance (i.e. a measured 8-hour urinary creatinine clearance >= 120 ml/min/1.73m²) in an adult non-critically ill abdominal and trauma surgery population.

Secondary objectives are the identification of risk factors associated with ARC in this specific study population.

In every included patient, an 8-hour urine collection was carried out over an 8-hour time period to determine the CrCl8h. Participants were asked to empty the bladder at the start of the collection. From then, patients were asked to collect urine in a recipient during the following 8 hours. If an indwelling transurethral or suprapubic urinary catheter was in situ, the collection bag was emptied at the start of the collection. After 8 hours, total urinary volumes (Uv8h) were measured with a measuring cup and urinary creatinine concentrations were determined by laboratory analysis (enzymatic analysis by Roche Diagnostics). Midterm serum creatinine samples were obtained at 4 hours after the start of the urinary collection. Based on these values, CrCl8h was calculated according to the standard formulas and normalized to a body surface area (BSA) of 1.73m².

The following demographic and clinical data were prospectively recorded or calculated: age, sex, total body weight, lean body weight, length, BMI, BSA, presence of an urinary catheter, pre- or postoperative status, 'preoperative American society of anesthesiology' (ASA) score, relevant medical history with respect to the kidney function or SCr levels (i.e. arterial hypertension, chronic kidney disease, diabetes mellitus, paralyzed patients or patients with amputated limb(s)), length of stay (LOS) since admission in the hospital until the day of collection (LOShosp), since admission on the ward until the day of collection (LOSward), since surgery until the day of collection (LOSsurgery), LOS in the hospital at discharge (LOSdisch), number of surgical interventions since admission until the day of collection, the mean daily volume of administered fluids based on the 3 days before the day of collection (d-3, d-2, d-1) as well as on the day of collection (d0), the relevant co-medication during d-3, d-2 and d-1 as well as d0, number of patients with one or more postoperative complication(s) (POC), number of POCs per patient and the highest severity grade of POCs per patient, C-reactive protein concentration (CRP) and white blood cell count (WBC) on d-1 or d0, baseline SCr (i.e. a SCr value from maximum 1 year old collected during a consultation), preoperative SCr (i.e. first SCr during hospital stay but before any surgical procedure) and SCr at discharge from the hospital. From the surgical procedure closest to the day of collection, we collected duration of anesthesia and surgical procedure, the administration of vasopressor agents, the volume and type of resuscitation fluids administered during surgery (i.e. crystalloids, colloids or blood derivates) and volumes of urine and blood loss. Additionally, in abdominal surgery patients, following demographic data were collected: elective or emergency surgical procedure, presence of a nasogastric tube and an ileo- or colostoma on the day of collection, reason for admission (i.e. colorectal, hepatobiliary or other), whether there was an oncologic indication for surgery and laparoscopic or open surgery. In trauma surgery patients following demographic data were collected additionally: the injury severity score (ISS) on admission, diagnosis at admission (i.e. trauma with fracture, trauma without fracture, infection, removal of osteosynthesis material or other) and type of fracture (if trauma with fracture). The type and severity of postoperative complications were classified using the Clavien-Dindo classification. All data were retrieved from the patient's computerized medical files and were registered in a patient study file (appendix 9.3) and in a Microsoft Office Access 2007 database.

ELIGIBILITY:
Inclusion Criteria:

* On the recruitment days, all non-critically ill adult patients hospitalized at the 74-bed abdominal and 50-bed trauma surgery wards in the 1850-bed University Hospitals Leuven were eligible for inclusion. On both wards, urinary collections are not routinely performed as part of standard of care.

Exclusion Criteria:

* Exclusion criteria were age younger than 18 years
* Do not resuscitate (DNR) code ≥ 2
* Discharge before 16 hour on the day of collection (d0)
* Surgery on the day of collection Pregnancy, lactation
* Renal replacement therapy
* Non-Caucasian ethnicity
* Isolation in order for source control due to infection with multi-drug resistant organisms (MDRO)
* Incontinence or the lack of cooperation
* At the abdominal ward in particular
* Women without an indwelling urinary catheter were also excluded due to the incapacity of these patients to carry out the urinary collection in a safe and painless manner
* During the urinary collection, patients with incomplete or doubtful urinary collections were excluded
* Patients could only be included once, except for those with incomplete urinary collection at an earlier day of collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of augmented renal clearance | 8 hours
  The prevalence of augmented renal clearance was calculated as the number of patients demonstrating a measured urinary creatinine clearnace ≥ 120 mL/min/1.73m² divided by the total number of included patients.

SECONDARY OUTCOMES:
Demographic and clinical factors independantly associated with augmented renal clearance | 6 months
  Demographic data, pre- or postoperative status, ASA score, relevant medical history with respect to the kidney function or SCr levels, interval from admission until the collection day, interval since surgery, LOS at discharge, number of surgical interventions, the mean daily volume of administered fluids based on the 3 days before the day of collection (d-3, d-2, d-1) as well as on the day of collection (d0), the relevant co-medication during d-3 until d0, patients with one or more postoperative complication (POC), number of POCs per patient and the highest severity grade of POCs per patient, CRP and white blood cell count (WBC) on d-1 or d0, baseline SCr, preoperative SCr and SCr at discharge from the hospital. From the surgical procedure closest to the day of collection, we collected duration of anesthesia and surgical procedure, the administration of vasopressor agents, the volume and type of resuscitation fluids administered during surgery and volumes of urine and blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Declercq, PharmD., Principal Investigator — Pharmacy Department, University Hospitals Leuven & Department of Pharmaceutical and Pharmacological Sciences, KULeuven, Belgium
Locations (1):
- Abdominal surgery ward and Trauma surgery ward, University Hospitals Leuven, Leuven, Vlaams Brabant, Belgium